CLINICAL TRIAL: NCT02250534
Title: Project 1, Study 2: Extended Exposure to Low Nicotine Content Cigarettes in Childbearing Age Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen T. Higgins, PhD, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: P50DA036114:P1S2; P50DA036114 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Tobacco Use Disorder
Keywords: Biomarkers of exposure; Compensatory smoking; Nicotine dependence; Reduced nicotine cigarettes; Tobacco withdrawal; Women; Health disparities; Vulnerable populations
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: This study was one of three multi-site clinical trials conducted in three different vulnerable populations under a similar protocol, with differences between protocols consisting of data collection specific to that vulnerable population. This included information such as use and timing of opioid maintenance therapy for individuals with opioid-use disorder or additional assessments of anxiety and depression for individuals with affective disorders. In order to explore potential differences across individuals with different vulnerabilities, data from all three studies were combined for analysis. A vulnerable population-by-condition or population-by- condition-by-time interaction term was included in all analyses. In the event that these interaction terms were statistically significant, all pairwise comparisons were conducted using a Bonferroni multiple comparison adjustment. Please see Statistical Analysis Plan for more details.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.8 mg nicotine (Experimental): 0.8 mg nicotine very low nicotine content cigarettes
  Interventions: Other: Very low nicotine content cigarettes
- 0.12 mg nicotine (Experimental): 0.12 mg nicotine very low nicotine content cigarettes
  Interventions: Other: Very low nicotine content cigarettes
- 0.03 mg nicotine (Experimental): 0.03 mg nicotine very low nicotine content cigarettes
  Interventions: Other: Very low nicotine content cigarettes

INTERVENTIONS:
Other: Very low nicotine content cigarettes

SUMMARY:
This study will examine extended exposure to cigarettes varying in nicotine content among disadvantaged women. Disadvantaged women are at increased risk for smoking, nicotine dependence, and using high nicotine yield cigarettes and are also at significantly increased risk for smoking-related adverse health consequences, including cervical cancer, thrombosis related to hormone-based contraception, infertility, and early menopause. Studies testing an innovative regulatory strategy of reducing the nicotine content of cigarettes to a non-addictive level have shown promising beneficial effects (decreased smoking rate, reduced toxicant exposure, and increased cessation) in the general population of smokers. However, these studies have uniformly excluded vulnerable populations like disadvantaged women who may respond differently considering their greater vulnerability to smoking and nicotine dependence. Thus, little is known scientifically about how this highly vulnerable subgroup of smokers might respond to a nicotine reduction policy. This project is designed to address that substantial knowledge gap. This same study was also conducted in two additional vulnerable populations under a similar protocol.

DETAILED DESCRIPTION:
The primary overall objective of these studies is to evaluate the effects of extended exposure to cigarettes differing in nicotine content in socioeconomically disadvantaged (< high school educational attainment) women of childbearing age using a 3-condition, parallel groups design. After a baseline period in which daily smoking rate and other baseline assessments are completed, participants will be randomly assigned to one of three cigarette conditions (nicotine content: 0.04, 2.4, and 15.8 mg nicotine/gram of tobacco) for the 12-week experimental period.

The cigarettes to be used in this study were made under an NIH contract with production being overseen by the Research Triangle Institute (referred to as "Spectrum cigarettes"). NIH currently has approximately 10 million of these cigarettes (of varying types) for research purposes. The cigarettes selected for the study span the range of yields likely to produce the hypothesized effects, as described above. The Spectrum cigarettes are not currently commercially available, although they are similar in many ways to marketed cigarettes (e.g., similar manufacturing, filter, paper, etc.).

The primary overall objective of this study is to evaluate the effects of extended exposure to cigarettes differing in nicotine content in female adult smokers of childbearing age (18-44 yrs) whose highest academic degree is high school using a 3-condition, parallel groups design. After a baseline period in which daily smoking rate and other baseline assessments are completed, participants will be randomly assigned to one of three cigarette conditions (nicotine content: 0.04 mg, 2.4 mg, and 15.8 mg nicotine/g of tobacco) for the 12-week experimental period.

Participants will be seen weekly throughout the 12-week experimental period to obtain research cigarettes. Cigarettes smoked per day will be obtained by participants completing daily Interactive Voice Response (IVR) reports of cigarettes in past 24 hours. This daily data will be used to calculate weekly means, with week-12 means serving as the primary outcome.

This same study was conducted in two additional vulnerable populations under a similar protocol, with differences between protocols consisting of data collection specific to that vulnerable population. This included information such as use and timing of opioid maintenance therapy for individuals with opioid-use disorder or additional assessments of anxiety and depression for individuals with affective disorders. In order to explore potential differences across individuals with different vulnerabilities, data from all three studies were combined for analysis. A vulnerable population-by-condition or population-by-condition-by-time interaction term was included in all analyses. In the event that these interaction terms were statistically significant, all pairwise comparisons were conducted using a Bonferroni multiple comparison adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-44 years
* Less than an Associate's degree
* Report smoking ≥ 5 cigarettes per day
* Provide an intake breath carbon monoxide (CO) sample > 8 ppm
* Be without current (within the past year) serious mental disorder that would interfere with study results or completion as determined by the Licensed Medical Professional or PI
* Be without current substance abuse/dependence other than nicotine
* Be sufficiently literate to complete research-related tasks
* Be in good physical health without serious illness or change in health or medication in the past three months as determined by the Licensed Medical Professional at each site
* Not pregnant or nursing and report using oral, implant, patch, ring, intrauterine device (IUD), injection, or barrier contraceptives or report being surgically sterile, or post menopausal
* Report no significant use of other tobacco or nicotine products within the past month (> 9 days in the past 30)

Exclusion Criteria:

* Any prior regular use (used as primary cigarette outside of the laboratory) of Spectrum cigarettes (i.e., research cigarettes with reduced nicotine content)
* Exclusive use of roll-your-own cigarettes
* Planning to quit smoking in the next 30 days
* A quit attempt in the past 30 days resulting in > 3 days of abstinence
* Currently taking anticonvulsant medications
* Positive toxicology screen for illicit drugs not including marijuana (participants with valid prescriptions will not be excluded and participants with a positive toxicology screen will be allowed to re-screen once)
* Breath alcohol level > 0.01 (participants with a positive screen will be allowed to re-screen once)
* Self-report of binge drinking alcohol (> 9 days in past 30, 4 drinks in 2 hours )
* Systolic blood pressure < 90 or ≥ 160 mmHg (participants outside the range will be allowed to re-screen once)
* Diastolic blood pressure < 50 or ≥ 100 mmHg (participants outside the range will be allowed to re-screen once)
* Breath CO > 80 ppm
* Heart rate < 45 or ≥ 115 bpm (participants outside the range will be allowed to re-screen once)
* Currently seeking treatment for smoking cessation
* Have used nicotine replacement, bupropion or other pharmacotherapies as cessation aids in the past month (bupropion for treatment of depression will be allowed)
* Current symptoms of psychosis, dementia or mania
* Suicidal ideation in the past month
* Suicide attempt in past 6 months
* Participation in another research study in the past 30 days

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 775 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T. Higgins, Ph.D., Study Director — University of Vermont; Sarah H. Heil, Ph.D., Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Harfmann RF, Heil SH, Bunn JY, Snell LM, Tidey JW, Sigmon SC, Gaalema DE, Lee DC, Streck JM, Bergeria CL, Davis DR, Plucinski S, Higgins ST. Changes in weight among individuals with psychiatric conditions or socioeconomic disadvantage assigned to smoke very low nicotine content cigarettes. Exp Clin Psychopharmacol. 2024 Apr;32(2):181-188. doi: 10.1037/pha0000700. Epub 2024 Jan 18. PMID 38236223
- [Derived] Gaalema DE, Snell LM, Tidey JW, Sigmon SC, Heil SH, Lee DC, Bunn JY, Park C, Hughes JR, Higgins ST. Potential effects of nicotine content in cigarettes on use of other substances. Prev Med. 2022 Dec;165(Pt B):107290. doi: 10.1016/j.ypmed.2022.107290. Epub 2022 Oct 5. PMID 36208817
- [Derived] Oliver AC, DeSarno M, Irvin CG, Kaminsky D, Tidey JW, Sigmon SC, Heil SH, Gaalema DE, Lee D, Bunn JY, Davis DR, Streck JM, Gallagher T, Higgins ST. Effects of Reduced Nicotine Content Cigarettes on Fractional Exhaled Nitric Oxide and Self-Reported Respiratory Health Outcomes Among Smokers With Psychiatric Conditions or Socioeconomic Disadvantage. Nicotine Tob Res. 2022 Jan 1;24(1):135-140. doi: 10.1093/ntr/ntab145. PMID 34255068
- [Derived] Higgins ST, DeSarno M, Bunn JY, Gaalema DE, Leventhal AM, Davis DR, Streck JM, Harfmann RF, Markesich C, Orr E, Sigmon SC, Heil SH, Tidey JW, Lee D, Hughes JR. Cumulative vulnerabilities as a potential moderator of response to reduced nicotine content cigarettes. Prev Med. 2021 Nov;152(Pt 2):106714. doi: 10.1016/j.ypmed.2021.106714. Epub 2021 Jul 7. PMID 34242666
- [Derived] Higgins ST, Tidey JW, Sigmon SC, Heil SH, Gaalema DE, Lee D, Hughes JR, Villanti AC, Bunn JY, Davis DR, Bergeria CL, Streck JM, Parker MA, Miller ME, DeSarno M, Priest JS, Cioe P, MacLeod D, Barrows A, Markesich C, Harfmann RF. Changes in Cigarette Consumption With Reduced Nicotine Content Cigarettes Among Smokers With Psychiatric Conditions or Socioeconomic Disadvantage: 3 Randomized Clinical Trials. JAMA Netw Open. 2020 Oct 1;3(10):e2019311. doi: 10.1001/jamanetworkopen.2020.19311. PMID 33079196
- [Derived] Higgins ST, DeSarno M, Davis DR, Nighbor T, Streck JM, Adise S, Harfmann R, Nesheim-Case R, Markesich C, Reed D, Tyndale RF, Gaalema DE, Heil SH, Sigmon SC, Tidey JW, Villanti AC, Lee D, Hughes JR, Bunn JY. Relating individual differences in nicotine dependence severity to underpinning motivational and pharmacological processes among smokers from vulnerable populations. Prev Med. 2020 Nov;140:106189. doi: 10.1016/j.ypmed.2020.106189. Epub 2020 Jul 3. PMID 32628945

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.8 mg Nicotine: 0.8 mg nicotine very low nicotine content cigarettes
  Very low nicotine content cigarettes
- 0.12 mg Nicotine: 0.12 mg nicotine very low nicotine content cigarettes
  Very low nicotine content cigarettes
- 0.03 mg Nicotine: 0.03 mg nicotine very low nicotine content cigarettes
  Very low nicotine content cigarettes
Period: Overall Study
Arm/Group | 0.8 mg Nicotine | 0.12 mg Nicotine | 0.03 mg Nicotine
Started | 254 | 235 | 286
Completed | 218 | 190 | 224
Not Completed | 36 | 45 | 62
Not completed — Lost to Follow-up | 18 | 28 | 33
Not completed — Personal reasons | 7 | 8 | 14
Not completed — Adverse Event | 6 | 3 | 8
Not completed — incarcerated | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Physician Decision | 1 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Reason unknown | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.8 mg Nicotine | 0.12 mg Nicotine | 0.03 mg Nicotine | Total
Number analyzed (Participants) | 254 | 235 | 286 | 775
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.90 (10.82) | 35.18 (11.13) | 35.65 (11.21) | 35.59 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 167 | 200 | 551
  Male | 70 | 68 | 86 | 224
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Latino White | 207 | 183 | 240 | 630
  Non-Latino Black | 24 | 25 | 19 | 68
  Latino | 7 | 8 | 8 | 23
  Non-Latino Other | 12 | 18 | 16 | 46
  Unknown | 4 | 1 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 254 | 235 | 286 | 775
Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes Per Day] | 19.63 (10.33) | 19.54 (10.56) | 19.91 (10.84) | 19.71 (10.58)

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day (CPD)
Description: Participant reported number of cigarettes smoked per day at Week 12.
Time Frame: 12 weeks
Population: Participants who completed Week 12.
Measure: Least Squares Mean (Standard Error); unit: cigarettes per day
Arm/Group | 0.8 mg Nicotine | 0.12 mg Nicotine | 0.03 mg Nicotine
Number analyzed (Participants) | 218 | 190 | 224
cigarettes per day | 25.28 (0.77) | 19.95 (0.80) | 17.74 (0.74)
Statistical Analysis 1: Comparison: 0.8 mg Nicotine vs 0.12 mg Nicotine; The statistical analysis method was ANCOVA, in order to test for statistically significant differences between group means, while controlling for covariates of interest. It was calculated that 207 subjects per group would be required to have at least 90% power to detect a mean difference of 4.52 CPD between the 0.8 mg and 0.12 mg groups at week 12, with significance level alpha of 0.0167. The significance level reflects the Bonferroni correction needed for testing of all pairwise comparisons; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is Bonferroni-corrected for multiple comparisons with a priori threshold of significance P < 0.0167; Mean Difference (Net) = -5.33, 95% CI 2-sided [-7.41 to -3.26], Standard Error of Mean 1.06 — Group difference = 0.12 mg nicotine - 0.8 mg nicotine
Statistical Analysis 2: Comparison: 0.8 mg Nicotine vs 0.03 mg Nicotine; The statistical analysis method was ANCOVA, in order to test for statistically significant differences between group means, while controlling for covariates of interest. It was calculated that 207 subjects per group would be required to have at least 90% power to detect a mean difference of 6.07 CPD between the 0.8 mg and 0.03 mg groups at week 12, with significance level alpha of 0.0167. The significance level reflects the Bonferroni correction needed for testing of all pairwise comparisons; Test type: Superiority; p < 0.0001, ANCOVA — The p-value is Bonferroni-corrected for multiple comparisons with a priori threshold of significance P < 0.0167; Mean Difference (Net) = -7.54, 95% CI 2-sided [-9.51 to -5.57], Standard Error of Mean 1.00 — Group difference = 0.03 mg nicotine - 0.8 mg nicotine

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | 0.8 mg Nicotine | 0.12 mg Nicotine | 0.03 mg Nicotine
All-Cause Mortality (participants affected / at risk) | 0/254 | 1/235 | 1/286
Serious Adverse Events (participants affected / at risk) | 13/254 | 4/235 | 13/286
Other Adverse Events (participants affected / at risk) | 241/254 | 203/235 | 226/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.8 mg Nicotine (N=254) | 0.12 mg Nicotine (N=235) | 0.03 mg Nicotine (N=286)
Sudden onset of chest pain due to not enough blood going to the heart (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bloody Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) — Diarrhea, Stomach pain, Vomiting
Kidney infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (2) — Cellulitis, Hepatitis B infection, Hepatitis C infection
Broken bone (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (7) — Bruising
Frontal lobe lesion (Investigations) | 0 (0) | 0 (0) | 1 (2) — Knee sprain
Diabetes Type 2 (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) — Hyperglycemia
Tenosynovitis of Hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (5) — Stroke
Anxiety, feelings of dread or danger (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) — Depression, Thoughts of taking ones own life
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin graft to wound on leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) — Hospitalization due to increased pain
High blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.8 mg Nicotine (N=254) | 0.12 mg Nicotine (N=235) | 0.03 mg Nicotine (N=286)
Infections and infestations (Infections and infestations) | 89 (113) | 79 (106) | 92 (119)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 78 (112) | 72 (111) | 84 (114)
Gastrointestinal disorders (Gastrointestinal disorders) | 63 (92) | 49 (71) | 77 (114)
General disorders (General disorders) | 58 (77) | 46 (72) | 67 (85)
Nervous system disorders (Nervous system disorders) | 49 (56) | 38 (52) | 46 (65)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 42 (52) | 27 (34) | 33 (41)
Vascular disorders (Vascular disorders) | 20 (30) | 22 (31) | 25 (34)
Surgical and medical procedures (Surgical and medical procedures) | 23 (28) | 16 (25) | 26 (31)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 22 (28) | 13 (13) | 17 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02250534/Prot_SAP_000.pdf